CLINICAL TRIAL: NCT03519828
Title: Effects of Oxidation-reduction Homeostasis on Cognitive Impairment in Patients With Ischemic Stroke
Brief Title: Oxidation-reduction Homeostasis in Cognitive Impairment Patients After Stroke
Status: Completed | Type: Observational
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Other Study IDs: k(2017)34
Record Dates: First submitted 2018-04-15; First posted 2018-05-09 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Oxidative-reduction Homeostasis; Post-stroke Cognitive Impairment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with post-stroke cognitive impairment
  Interventions: Other: No intervention has been conducted
- Patients without post-stroke cognitive impairment
  Interventions: Other: No intervention has been conducted

INTERVENTIONS:
Other: No intervention has been conducted — It is an observational study, and no intervention has been conducted

SUMMARY:
Cognitive impairment after ischemic stroke can affect not only the social adaptation ability, but also affect the comprehensive rehabilitation of patients. The damage of cognitive impairment after ischemic stroke is not lower than the body function defect after stroke. Many studies have shown that oxidative stress is one of the pathophysiological mechanisms of ischemic cerebrovascular disease. Many studies have reported that the oxidative-reduction of cells plays an important role in the life activities of organisms, affecting the health, aging and death of the organism. In the recent years, some scholars have suggested that post-stroke cognitive impairment may be related to oxidative-reduction homeostasis of the body, but the relevant evidence is lacking and needs to be further explored. Therefore, the purpose of this study is to explore the effect of oxidation-reduction homeostasis on cognitive impairment in patients with ischemic stroke, and provide a theoretical basis for the prevention and treatment of cognitive impairment after ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years old;
* Ischemic stroke for the first time or previous stroke but with no serious sequelae (mRS is 0 -2 points);
* Time from onset to treatment ≤48 hours;
* Conscious awareness, and with no obvious aphasia and visual impairment;
* Signed informed consent by patient self or legally authorized representatives.

Exclusion Criteria:

* Intracranial hemorrhage or suspected subarachnoid hemorrhage;
* Transient ischemic attack;
* Patients with severe mental disorders or language disorders;
* Patients can not cooperate with evaluators, such as mental illness or dementia;
* Pregnant women or suckers;
* Researchers consider patients inappropriate to participate in the registry.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients in hospital from March, 2018 to September, 2018.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Oxidative-reduction homeostasis in acute ischemic stroke patients | 1 day
  Reduced glutathione (GSH)/ Oxidized glutathione (GSSG), Superoxide dismutase (SOD), Catalase (CAT), Glutathione Peroxidase (GSH-PX) of acute ischemic stroke patients will be tested.
Cognitive function in acute ischemic stroke patients | 1 day
  Mini Mental Status Examination (MMSE) and Montreal cognitive assessment scale (MoCA) in acute ischemic stroke patients will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No